CLINICAL TRIAL: NCT03135808
Title: Surgical Anatomy and 'Waisting' of the sIgmoid SpEcimen
Acronym: WISE
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Pelican Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4686
Record Dates: First submitted 2017-04-05; First posted 2017-05-01 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Sigmoid, Sigmoid Colon, Neoplasm, Cancer
Keywords: MRI; Imaging,; Anatomy; Tissue; Colorectal; Sigmoid; Colon; Pathology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Treatment of rectal cancer has improved to the extent that its local recurrence rates are now much lower than other sites in the large bowel. It has been found that higher rates of recurrence in the sigmoid section of the colon, just before the rectum. This might be due to a narrowing in the bowel, and difficulties identifying whether cancers are in the sigmoid or rectum. The aim is to investigate the bowel from 20 patients undergoing surgery for left sided colorectal cancer at the Royal Marsden. These patients would have routine investigations and treatments, but once the bowel has been removed, it would undergo a MRI scan and additional slices and photography during pathological analysis.

DETAILED DESCRIPTION:
Following surgery for a primary cancer (ie has not spread), the patient may still die from the cancer. This may be due to local or distant recurrence. Local recurrence will be near the site of the surgery; for bowel cancer, this may be at the site of the joined bowel or nearby in the abdomen. Distant recurrence will be elsewhere in the body.

Local recurrence is much more likely when there is incomplete removal of all the cancer cells at the time of surgery This can occur if the surrounding tissue, such as the bowel mesentery, is not completely removed. The bowel mesentery is the fatty tissue in which blood vessels and lymph nodes travel up to the bowel. During research into rectal cancer, it was established that there was a rectal mesentery "waist" or narrowing that made it difficult with conventional surgery to remove all the cancer cells. A modified operation gave much better cancer clearance.

Rectal cancer outcomes are now superior to other sites of large bowel cancer. Data from the Royal Marsden and elsewhere show that local recurrence rates of the sigmoid colon are approximately double that of the rectum. This may be due to 2 potential issues: a sigmoid waist, and difficulties in differentiating rectal and sigmoid cancers.

This recurrence may be due to the presence of a waist in the sigmoid mesentery. A case series from Leeds has shown initial data suggesting there is a significantly smaller area in this area. However, this study was underpowered and not conducted prospectively in a scientifically rigorous manner. If a waist was present that could prevent cancer being successfully removed, then an extended operation could be performed or radiotherapy/chemotherapy given before the operation to shrink the cancer.

The sigmoid colon is the section of bowel before the rectum. They can be differentiated by examining the bowel during or after the operation for specific landmarks (taenia coli, appendices epiploicae) that are present on the sigmoid but not on the rectum. However, these landmarks cannot be seen on a patient's pre-operative scans, making it is very difficult to tell whether a cancer is in the sigmoid or the rectum. At our institution, we use MRI to define the end of the sigmoid at MRI as the transition point from the sigmoid mesocolon to the mesorectal apex. This can be seen on sagittal views between the fanning branches of the sigmoid artery proximally and the superior rectal vein distally. On axial views, it can be seen when the rectum fixed posteriorly by the mesorectum transitions into the sigmoid hanging freely on the sigmoid mesocolon. If the distance from the anterior peritoneal reflection to the mesorectal apex on MRI or the coalescence of the taenia coli on histology correlate, it can be predicted pre-operatively on MRI whether a patient's cancer is in the sigmoid or the rectum, and what kind of treatment they should undergo.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years with rectal or sigmoid cancer who will be undergoing left sided colorectal resection including the anterior peritoneal reflection.
* Patients must be able to undergo colonoscopy, adequate bowel preparation, MRI and surgery.

Exclusion Criteria:

* Patients who are unable to consent, withhold consent or withdraw consent, including patients who require an emergency operation and will be unable to give informed consent
* Contraindication to MRI as per MHRA recommendations [36] eg implanted medical devices, severe claustrophobia
* Distortion of the sigmoid mesentery due to tumour perforation, invasion (stage T4), or extreme bulk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 years with rectal or sigmoid cancer who will be undergoing left sided colorectal resection including the anterior peritoneal reflection.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Height from peritoneal reflection to the mesorectal apex in mm, from the pathology specimen. | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross sectional slices using a high definition camera and will be used to perform the necessary measurements for the study.
The area of tissue in mm2 within the mesentery, from the pathology specimen. | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross

SECONDARY OUTCOMES:
Distance in mm from the anterior peritoneal reflection to the rectosigmoid junction on MRI (mesorectal apex, insertion of the superior rectal artery, sacral promontory, inferior border of S2) vs pathology specimen (coalescence of taenia coli). | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross sectional slices using a high definition camera and will be used to perform the necessary measurements for the study.
Height from peritoneal reflection to the mesorectal apex in mm, on MRI vs pathology specimen. | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross sectional slices using a high definition camera and will be used to perform the necessary measurements for the study.
The area in mm2 of tissue within the mesentery, on MRI vs pathology specimen. | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross sectional slices using a high definition camera and will be used to perform the necessary measurements for the study.
Height from peritoneal reflection to the mesorectal apex in mm by location (anterior, posterior, left and right lateral), on MRI vs pathology specimen. | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross sectional slices using a high definition camera and will be used to perform the necessary measurements for the study.
The area of tissue in mm2 within the mesentery by location (anterior, posterior, left and right lateral), on MRI vs pathology specimen. | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross sectional slices using a high definition camera and will be used to perform the necessary measurements for the study.
Height from peritoneal reflection to the mesorectal apex in mm, by compass direction, on MRI vs pathology specimen. | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross sectional slices using a high definition camera and will be used to perform the necessary measurements for the study.
The diameter in mm of tissue within the mesentery by compass direction, on MRI vs pathology specimen. | 48 hours post-surgery
  Photographs will be captured of the macroscopic whole specimen and serial cross sectional slices using a high definition camera and will be used to perform the necessary measurements for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, Principal Investigator — Consultant Radiologist and Professor in Cancer Imaging
Locations (1):
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No